CLINICAL TRIAL: NCT04130074
Title: Role of Duplex Doppler In Diagnosis of Acute Appendicitis : in Correlation With Surgical Management Outcome
Brief Title: Role of Duplex Doppler in Accurate Diagnosis of Appendicitis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: abdelRahman Ahmad abdAllah (Other)
Responsible Party: Sponsor-Investigator, abdelRahman Ahmad abdAllah, resident doctor, Assiut University
Organization: Assiut University (Other)
Other Study IDs: US in appendecitis
Record Dates: First submitted 2019-10-15; First posted 2019-10-17 (Actual); Last update posted 2020-06-05 (Actual); Status verified 2020-06

CONDITIONS: Appendicitis Acute
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

INTERVENTIONS:
Device: duplex doppler ultra sound and CT — graded compression US done in different positions then take MSCT with contrast on abdomen to compare with

SUMMARY:
To evaluate the role of duplex doppler in diagnosis of appendicitis compared to CT

DETAILED DESCRIPTION:
Acute appendicitis (AA) is the most common acute abdominal condition worldwide [1]

Thus far, the clinical diagnosis of (AA) remains a challenge to emergency physicians and surgeons both in the pediatric and adult populations, as the symptoms are often atypical and overlapped with various other diseases[2],[3].

The accurate diagnosis of AA depends on both clinical presentations and imaging techniques.

To date, US and computed tomography (CT) remain the most common used diagnostic imaging, and CT is considered the gold standard technique to evaluate patients with suspected AA, because of its high sensitivity and specificity [2],[3]. While the associated radiation exposure remains a concern, especially, among children, the elderly and pregnant women, as radiation protection is of major importance [2],[3],[5],[6].

Over recent years, research on various aspects of US imaging in the diagnosis of (AA) has gained major importance due to its radiation protection, broad availability and cost-effectiveness [6].

Therefore,US may be valuable as an initial imaging choice for patients with suspected (AA) or with equivocal clinical presentations [7],[8].

With continuing efforts to improve the diagnostic performance of US, a variety of US findings have been described for use in the setting of suspected appendicitis, including the maximum outer diameter (MOD), periappendiceal fluid, echogenic periappendiceal fat, and loss of the normally echogenic submucosal layer within the appendiceal wall [9] ,[10].

Color Doppler imaging has been utilized as well, with early reports describing no detectable flow in the normal appendix and later reports, with the benefit of improved instrumentation, d describing flow in normal appendices and hyperemia in inflamed appendices [11],[12].

However, objective criteria for interpreting Doppler results generally have not been specifically described [11],[13],[12],[14].

.Spectral Doppler imaging, in contrast to color Doppler imaging, provides inherently objective, quantitative data such as peak systolic velocity (PSV) and resistive index (RI) values. These measurements have found utility in the assessment of the carotid arteries and, for example, both native as well as transplanted hepatic and renal vessels[16],[17]. Early investigations addressed the RI in appendicitis as well, without emphasis on the PSV, using instrumentation that was modern for the time [18],[19],[20].

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute abdomen and suspected appendicitis.

Exclusion Criteria:

* so Obese and irritable Patients whom satisfactory graded compression US can't be done.
* pregnant women , children under 3 years old and adults over 60 years old for radiation hazards.
* patients with renal impairment for contrast hazards.

Ages: 3 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients with acute abdomen and suspected appendicitis.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-07-05 (Estimated); Primary Completion 2021-02-15 (Estimated); Study Completion 2021-03-15 (Estimated)

PRIMARY OUTCOMES:
comparison of duplex Doppler results with CT results | baseline
  PSV = peak systolic velocity in cm/second , PDV =peak diastolic velocity in cm/second, and PI =( PSV - PDV)/ PSV taken from the intra mural appendiceal artery then compare with the results of MSCT with contrast of the abdomen.

CONTACTS AND LOCATIONS:
Locations (1):
- Diagnostic Radiology Department of the assiut university hospital, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blitman NM, Anwar M, Brady KB, Taragin BH, Freeman K. Value of Focused Appendicitis Ultrasound and Alvarado Score in Predicting Appendicitis in Children: Can We Reduce the Use of CT? AJR Am J Roentgenol. 2015 Jun;204(6):W707-12. doi: 10.2214/AJR.14.13212. PMID 26001260
- [Background] Humes DJ, Simpson J. Acute appendicitis. BMJ. 2006 Sep 9;333(7567):530-4. doi: 10.1136/bmj.38940.664363.AE. No abstract available. PMID 16960208
- [Background] Shogilev DJ, Duus N, Odom SR, Shapiro NI. Diagnosing appendicitis: evidence-based review of the diagnostic approach in 2014. West J Emerg Med. 2014 Nov;15(7):859-71. doi: 10.5811/westjem.2014.9.21568. Epub 2014 Oct 7. PMID 25493136
- [Background] Mostbeck G, Adam EJ, Nielsen MB, Claudon M, Clevert D, Nicolau C, Nyhsen C, Owens CM. How to diagnose acute appendicitis: ultrasound first. Insights Imaging. 2016 Apr;7(2):255-63. doi: 10.1007/s13244-016-0469-6. Epub 2016 Feb 16. PMID 26883138
- [Background] Brenner D, Elliston C, Hall E, Berdon W. Estimated risks of radiation-induced fatal cancer from pediatric CT. AJR Am J Roentgenol. 2001 Feb;176(2):289-96. doi: 10.2214/ajr.176.2.1760289. PMID 11159059
- [Background] Hernandez JA, Swischuk LE, Angel CA, Chung D, Chandler R, Lee S. Imaging of acute appendicitis: US as the primary imaging modality. Pediatr Radiol. 2005 Apr;35(4):392-5. doi: 10.1007/s00247-004-1372-8. Epub 2005 Jan 6. PMID 15635471
- [Background] Rice HE, Arbesman M, Martin DJ, Brown RL, Gollin G, Gilbert JC, Caty MG, Glick PL, Azizkhan RG. Does early ultrasonography affect management of pediatric appendicitis? A prospective analysis. J Pediatr Surg. 1999 May;34(5):754-8; discussion 758-9. doi: 10.1016/s0022-3468(99)90369-x. PMID 10359177
- [Background] Chan L, Shin LK, Pai RK, Jeffrey RB. Pathologic continuum of acute appendicitis: sonographic findings and clinical management implications. Ultrasound Q. 2011 Jun;27(2):71-9. doi: 10.1097/RUQ.0b013e31821b6eea. PMID 21606789
- [Background] Trout AT, Towbin AJ, Fierke SR, Zhang B, Larson DB. Appendiceal diameter as a predictor of appendicitis in children: improved diagnosis with three diagnostic categories derived from a logistic predictive model. Eur Radiol. 2015 Aug;25(8):2231-8. doi: 10.1007/s00330-015-3639-x. Epub 2015 Apr 28. PMID 25916384
- [Background] Ohba G, Hirobe S, Komori K. The Usefulness of Combined B Mode and Doppler Ultrasonography to Guide Treatment of Appendicitis. Eur J Pediatr Surg. 2016 Dec;26(6):533-536. doi: 10.1055/s-0035-1570756. Epub 2016 Jan 8. PMID 26745520
- [Background] Gaitini D, Beck-Razi N, Mor-Yosef D, Fischer D, Ben Itzhak O, Krausz MM, Engel A. Diagnosing acute appendicitis in adults: accuracy of color Doppler sonography and MDCT compared with surgery and clinical follow-up. AJR Am J Roentgenol. 2008 May;190(5):1300-6. doi: 10.2214/AJR.07.2955. PMID 18430847
- [Background] Kessler N, Cyteval C, Gallix B, Lesnik A, Blayac PM, Pujol J, Bruel JM, Taourel P. Appendicitis: evaluation of sensitivity, specificity, and predictive values of US, Doppler US, and laboratory findings. Radiology. 2004 Feb;230(2):472-8. doi: 10.1148/radiol.2302021520. Epub 2003 Dec 19. PMID 14688403
- [Background] Linam LE, Munden M. Sonography as the first line of evaluation in children with suspected acute appendicitis. J Ultrasound Med. 2012 Aug;31(8):1153-7. doi: 10.7863/jum.2012.31.8.1153. No abstract available. PMID 22837278
- [Background] Baldisserotto M, Peletti AB. Is colour Doppler sonography a good method to differentiate normal and abnormal appendices in children? Clin Radiol. 2007 Apr;62(4):365-9. doi: 10.1016/j.crad.2006.11.009. Epub 2007 Jan 30. PMID 17331831